CLINICAL TRIAL: NCT00042900
Title: A Phase I Clinical And Pharmacological Study Of Pyroxamide (NSC 696085) In Patients With Advanced Malignancies
Brief Title: Pyroxamide in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 99-090; CDR0000069483 (Registry Identifier: PDQ (Physician Data Query)); NCI-2110
Record Dates: First submitted 2002-08-05; First posted 2003-07-08 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous Condition; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; T-cell large granular lymphocyte leukemia; Waldenström macroglobulinemia; accelerated phase chronic myelogenous leukemia; acute undifferentiated leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; primary myelofibrosis; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; essential thrombocythemia; extramedullary plasmacytoma; intraocular lymphoma; isolated plasmacytoma of bone; meningeal chronic myelogenous leukemia; monoclonal gammopathy of undetermined significance; polycythemia vera; previously treated myelodysplastic syndromes; primary central nervous system non-Hodgkin lymphoma; primary systemic amyloidosis; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; small intestine lymphoma; stage III adult Hodgkin lymphoma; stage III adult T-cell leukemia/lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III cutaneous T-cell non-Hodgkin lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III multiple myeloma; stage III mycosis fungoides/Sezary syndrome; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV chronic lymphocytic leukemia; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV mycosis fungoides/Sezary syndrome; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated hairy cell leukemia; stage IV adult Hodgkin lymphoma; stage IV adult T-cell leukemia/lymphoma; unspecified adult solid tumor, protocol specific; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Primary Myelofibrosis; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Thrombocythemia, Essential; Intraocular Lymphoma; Monoclonal Gammopathy of Undetermined Significance; Polycythemia Vera; Immunoglobulin Light-chain Amyloidosis; Leukemia, Prolymphocytic; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Lymphoma, B-Cell, Marginal Zone | interventions — pyroxamide

INTERVENTIONS:
Drug: pyroxamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of pyroxamide in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of pyroxamide in patients with advanced malignancies.
* Define, qualitatively and quantitatively, the dose-limiting and non-dose-limiting toxic effects of this drug in these patients.
* Describe the pharmacologic behavior of this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive pyroxamide IV continuously over 5-7 days. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of pyroxamide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for resolution of adverse events.

PROJECTED ACCRUAL: A maximum of 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor or hematologic malignancy

  * Disease that has failed standard therapies (e.g., surgery, radiotherapy, endocrine therapy, or chemotherapy) or for which no curative or life- prolonging therapy is available
* Measurable or clinically evaluable disease

  * Elevated tumor marker is acceptable for evaluable disease
* No known carcinomatous meningitis, primary brain tumors, or metastatic brain disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 125,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* Bilirubin normal
* AST no greater than 2.5 times upper limit of normal (ULN) (5 times ULN if liver metastases present)
* PT no greater than 1.5 times ULN

Renal

* Creatinine normal

Other

* HIV-positive status allowed
* Prior malignancy allowed
* No severe physical or emotional illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent bone marrow growth factors

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* At least 4 weeks since prior wide-field radiotherapy and recovered
* At least 2 weeks since prior limited-field radiotherapy and recovered
* Recovered from prior radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent antitumor treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard B. Saltz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States